CLINICAL TRIAL: NCT04762732
Title: The Use of Incisional Negative Pressure Wound Therapy for Management of Anterolateral Thigh Flap Donor Site Wound: A Prospective, Randomized Controlled Study
Brief Title: The Use of iNPWT for Management of ALT Flap Donor Site Wound
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202006043RIPD
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Incisional Negative Pressure Wound Therapy
Keywords: free flap, head and neck cancer, wound care
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: negative pressure wound therapy(PREVENA™ Incision Management System) (Experimental): Wound of ALT donor site will be cared under PREVENA™ Incision Management System
  Interventions: Device: NPWT
- Placebo Comparator: conventional dressing (Placebo Comparator): Wound of ALT donor site will be cared by traditional dressing and care.
  Interventions: Device: Traditional wound care

INTERVENTIONS:
Device: NPWT — Wound of ALT donor site will be cared under PREVENA™ Incision Management System for 5 days post-operatively.
  Arms: Experimental: negative pressure wound therapy(PREVENA™ Incision Management System)
Device: Traditional wound care — Wound of ALT donor site will be covered by vaseline gauze coated with tetracycline ointment (Genuine Chemical Pharmaceutical, Tao-Yuan, Taiwan), and layers of gauze.
  Arms: Placebo Comparator: conventional dressing

SUMMARY:
Primary closure or skin grafting of the donor site after harvest of a anterolateral thigh flap (ALT) is associated with significant morbidity. Incisional negative pressure wound therapy (NPWT) may decrease complications in high-risk incisions. Successful use of NPWT has been reported in the treatment of ALT flap donor site wounds in a retrospective observational study, but no prospective study of NPWT application in the ALT flap donor site has been reported. This study aims to assess the incidence of complications at ALT flap donor site with an incisional NPWT device, PREVENA™. A prospective, controlled, pair-matched study has been designed to compare the effectiveness, complication rate, and scar quality of ALT flap donor site between using incisional NPWT and conventional bolster dressing.

DETAILED DESCRIPTION:
Primary closure or skin grafting of the donor site after harvest of a anterolateral thigh flap (ALT) is associated with significant morbidity. Incisional negative pressure wound therapy (NPWT) may decrease complications in high-risk incisions. Successful use of NPWT has been reported in the treatment of ALT flap donor site wounds in a retrospective observational study, but no prospective study of NPWT application in the ALT flap donor site has been reported. This study aims to assessed the incidence of complications at ALT flap donor site with an incisional NPWT device, PREVENA™. A prospective, controlled, pair-matched study has been designed to compare the effectiveness, complication rate, and scar quality of ALT flap donor site between using incisional NPWT and conventional bolster dressing.

ELIGIBILITY:
The study is designed as a prospective randomized clinical trial. This study aims to enroll patients who require a free ALT flap for head and neck reconstruction. Inclusion criteria are as follows:

1. The donor site of ALT flap can be closed primarily.
2. Age≥20 years and <80 years
3. ALT flap size measuring more than 6 cm in width
4. Patients will be required to understand and be willing to participate in the trial and be able to comply with the follow-up visits

Exclusion criteria are as follows:

1. he donor site of ALT flap can not be closed primarily.
2. Uncontrolled diabetes mellitus, as measured by HbA1c≥10%
3. Under renal replacement therapy for more than 1 year.
4. Pregnant woman

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Development of wound dehiscence or other wound complications in the ALT flap donor site area | 30 days
  Development of wound dehiscence or other wound complications in the ALT flap donor site area during the first 6 weeks postoperatively. Wound dehiscence is defined as the splitting apart or rupturing of the margins of a previously closed wound along some or all of its length. Surgical site infection (SSI) was reported according to the revised criteria outlined by the Centers for Disease Control and Prevention (CDC), USA. To achieve a higher degree of objectivity, we will also adopt the modified ASEPSIS score criteria and definitions. The primary outcomes are assessed at the standardized follow-up visits by nurses and physicians in the hospital or in the outpatient clinic, who are not connected to the study and blinded to dressing allocation. The presence of dehiscence/infection at the ALT flap donor site, total or partial skin graft loss, and the need for another surgical procedure to the donor site are recorded.

SECONDARY OUTCOMES:
donor site scar quality | 6 months
  irst, we will use the Vancouver Scar Scale (VSS) for evaluation at post-operative 6 months. The VSS assesses four variables: vascularity, height/thickness, pliability and pigmentation. Each variable includes ranked subscales that are summed to obtain a total score ranging from 0 to 13, with 0 representing normal skin and 13 representing maximum alterations of the skin. The Patient and Observer Scar Assessment Scale (POSAS), which is a reliable and consistent tool used to assess scar quality, will also be employed.

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Chen Cheng, PhD, Principal Investigator — Division of Plastic Surgery, Department of Surgery, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan